CLINICAL TRIAL: NCT05374044
Title: Establishment of a Quantified Imaging Method for Evaluating Tumor Response Grade in Rectal Cancer Patient With Neoadjuvant Therapy: a Multi-center Study
Brief Title: Establishment of MRI Model for pTRG in Rectal Cancer With Establishment of
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Capital's Funds for Health Improvement and Research (2020-1- 2151). (Unknown)
Responsible Party: Principal Investigator, Sun Ying-Shi, Professor, Peking University Cancer Hospital & Institute
Other Study IDs: SF2020-1-2151
Record Dates: First submitted 2021-12-14; First posted 2022-05-13 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; neoadjuvant therapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- rectal cancer with NAT: The patients are planned to receive neoadjvant therapy, and then receive radical surgery.
  Interventions: Diagnostic Test: pelvic MRI for establishing new mrTRG method

INTERVENTIONS:
Diagnostic Test: pelvic MRI for establishing new mrTRG method — they will received two pelvic MR examinations before and after neoadjvant therapy. The MRI before neoadjvant therapy is considered as baseline MRI, which is usually taken within 3 weeks before NAT. The MRI after neoadjvant therapy is considered as preoperative MRI, which is usually taken within 3-8 weeks before NAT.

SUMMARY:
This study proposeto integrate a variety of imaging quantitative indicators to establish a new MRI-based tumor response regression(mrTRG) classification method. The accuracy of the established mrTRG classification method according pathology TRG(pTRG) will be tested. The ability of the established mrTRG classification method to predict prognosis will also be tested.

DETAILED DESCRIPTION:
The study included two part: one is a retrospective single-center cohort for analyzing quantitative MRI factors associated with pTRG, from which a new MRI-based tumor response regression(mrTRG) classification method will be established. The other is a prospective multi-center cohort for testing the accuracy of the established mrTRG classification according to pTRG; and also for validating the established mrTRG classification associated with survival.

ELIGIBILITY:
Inclusion Criteria:

* biopsy-proved primary rectal cancer
* baseline MRI confirmed LARC (cT3 and/or cN+)
* scheduled to take neoadjuvant therapy
* receive baseline and preoperative pelvic MRI
* receive TME surgery after NAT
* have routine follow-up after the operation

Exclusion Criteria:

* history of malignancy or multiple primary cancers
* receive surgery directly without NAT
* don't receive TME surgery
* don't complete NAT
* simultaneous distant metastasis at the baseline diagnosis
* lack of baseline or preoperative pelvic MRI
* incomplete or unavailable pathological information
* lost to follow-up within three months after surgery (lost since the first follow-up visit)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: biopsy-proved primary locally advanced rectal adenocarcinoma(cT3 and/or cN+)
Sampling Method: Probability Sample
Enrollment: 385 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
pathological tumor regression grade(pTRG) | within 2 weeks after surgery
  pTRG is evaluated according to the AJCC system. pTRG0-1 is defined as good response, pTRG2 as moderate response, and pTRG3 as poor response. The pTRG is judged by two experienced pathologists working together. If there are any discrepancies, then a third senior pathologist is consulted for arbitration. there were any discrepancies, then a third senior pathologist was consulted. there were any discrepancies, then a third senior pathologist was consulted.

SECONDARY OUTCOMES:
distant metastasis | 3 years from the data of surgery
  Distant metastastic lesion detected by follow-up CT which will be performed every 3 month for the first two year and every 6 month since the third year
Death | 3 years from the data of surgery
  all cause death
local recurrence | 3 years from the data of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Shi Sun, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (3):
- China (3):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking University Shougang Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Undecided